CLINICAL TRIAL: NCT03312673
Title: Asthma, Smoking, Emotional Deficits
Acronym: ASTADEM
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0159
Record Dates: First submitted 2017-10-04; First posted 2017-10-18 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Asthma; Emotional Disorder; Alexithymia
MeSH Terms: conditions — Asthma; Affective Symptoms | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Asthma population: Patients (men and women) asthmatic smokers and non-smokers followed routinely in the pulmonology department, Croix-Rousse Hospital, Hospices Civils of Lyon.
  Interventions: Other: Interview and tests of drawing.

INTERVENTIONS:
Other: Interview and tests of drawing. — The intervention will take place with patients followed for asthma at the Croix Rousse hospital. Patients agreeing to participate in the study will come to the hospital for one hour and a half. They will answer questionnaires and tests of drawing. Results Restitution Session (optional) is proposed to patients within the next 4 weeks during a routine consultation.

SUMMARY:
The objective of the study is to determine whether poor control of asthma is related to an emotional deficit such as alexithymia. The hypothesis is that there is a correlation between the severity of asthma, its control, and the degree of emotional deficits.

ELIGIBILITY:
Inclusion Criteria:

* Men and women (> 18 years).
* Asthma (mild, moderate, severe).
* Beneficiary of social security

Exclusion Criteria:

* Pregnant women
* Patients who oppose their participation in the study
* Multiple drug users (psychoactive substances).
* Patients with severe psychiatric antecedents and comorbidities.
* Patients with cancer
* Patients with cognitive impairment
* Patients with speech, hearing, visual, and praxic disorders.
* Any chronic and especially respiratory pathology other than asthma (COPD, bronchiectasis), which can alter the study.
* Patients not speaking French
* Persons protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asthma sufferers treated at the Croix Rousse hospital
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
Poor control of asthma | During routine visit (one hour and a half)
  The poor asthma control is defined by a score <20 on the ACT test
Emotional deficit such as alexithymia | During routine visit (one hour and a half)
  Defined by a score ≥ 44 points/100 on the Toronto scale
Emotional deficit indicator traces | During routine visit (one hour and a half)
  Identifying indicator traces of emotional deficits according to the dimensions defining the alexithymia on the test of the tree and the drawing of the person
Depression | During routine visit (one hour and a half)
  Defined by a score ≥ 11 points on the HADS scale
Anxiety | During routine visit (one hour and a half)
  Defined by a score ≥ 11 points on the HADS scale
Emotional valences | During routine visit (one hour and a half)
  Defined by 8 scores distinct on Diener's subjective well-being scale

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Pneumologie Hôpital de la Croix-Rousse, Lyon, France

IPD SHARING:
Plan to Share IPD: No